CLINICAL TRIAL: NCT01010685
Title: Safety and Feasibility Trial of Laparoscopic Small Port Cholecystectomy With Transgastric Gallbladder Recovery
Brief Title: Safety Study of Keyhole Gallbladder Surgery With Removal of Gallbladder Via the Stomach Rather Than Through the Skin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Specialised equipment required withdrawn from market
Sponsor: Colchester Hospital University NHS Foundation Trust (Other Government)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Mr Ralph Austin, Consultant laparoscopic surgeon, Colchester Hospital University NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0302/104
Record Dates: First submitted 2009-11-07; First posted 2009-11-10 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Gallstones
Keywords: Natural Orifice Transluminal Endoscopic Surgery (NOTES); Transgastric surgery; Surgical Procedures, Minimally Invasive
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Recovery of gallbladder via gastrotomy instead of via the skin — The gallbladder is dissected as for a standard laparoscopic cholecystectomy but is then recovered via a hole in the stomach created and closed endoscopically rather than through the skin as in the standard fashion

SUMMARY:
The benefits of laparoscopic ("minimally invasive" or "keyhole") surgery for gallbladder removal (cholecystectomy) over open surgical procedures in terms of significant reductions in pain, scarring and recovery time are well accepted. In a conventional laparoscopic cholecystectomy however, the excised gallbladder still has to be extracted through the abdominal wall skin via a laparoscopic port site using an incision of 10mm or greater. Despite being much smaller than that required for open surgery, this incision is painful, leaves a scar and can result in a port site hernia to follow requiring further surgery to repair it. Recent attempts to further reduce the invasiveness of the surgical procedure have suggested performing the operation via an endoscope passed through the mouth and through an incision in the stomach wall - so called Natural Orifice Translumenal Endoscopic Surgery (NOTES). Unlike a skin incision, an incision in the wall of the stomach (gastrotomy) should give no pain, visible scar or herniation risk yet still allow access to the peritoneal cavity for surgical procedures such as cholecystectomy. Against this, it has the potential risks of contamination and leakage of gastric contents into the peritoneal cavity. Whilst the limitations of present technology make it very difficult to perform an entire cholecystectomy through the stomach wall in patients, endoscopic methods for closing a gastrotomy are available that are approved for use in patients (CE marked) and it is hypothesised that removing the excised gallbladder through the stomach in this way would avoid the problems of extracting it through the abdominal wall described above. Data are required to determine whether the extraction of the gallbladder via a gastrotomy rather than through the skin is safe, producing smaller scars and a better cosmetic result. A secondary endpoint would be to assess possible reductions in pain and recovery from this less invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Fit patients, avoiding extremes of age, with uncomplicated gallstone disease requiring elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Direct healthcare team deny permission to approach patient for trial.
* Patient request / preference.
* Age (< 21 or > 65 yrs old).
* Co-morbidity (ASA level 3 or above).
* BMI > 32.
* Complicated gallstone disease (eg bile duct stones/ERCP/pancreatitis).
* Gallstones ≥ 18 mm size (too large to recover via oesophagus).
* Pregnancy.
* Previous gastric or upper abdominal surgery (alterations in gastric anatomy or adhesions preventing safe gastrotomy).
* Emergency procedure.
* Planned other operation during cholecystectomy.
* Inability to consent or psychiatric or addiction problems relevant to surgery.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
This is a pilot study aimed at examining the outcomes of gallbladder recovery through a gastrotomy, concentrating on safety. The main outcome is presence of surgical complications. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes include pain levels and cosmetic satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Austin, MS, FRCS, Principal Investigator — Colchester General Hospital
Locations (1):
- Colchester General Hospital, Colchester, Essex, United Kingdom